CLINICAL TRIAL: NCT03723395
Title: A Phase 1, Open-Label, Fixed-sequence, 5-part, Drug-drug Interaction Study of Tucatinib to Evaluate the Effects of CYP3A4 and CYP2C8 Inhibition and Induction on the Pharmacokinetics of Tucatinib and to Evaluate the Effects of Tucatinib on the Pharmacokinetics of Substrates of CYP3A4, CYP2C8, CYP2C9, and P-glycoprotein in Healthy Male and Female Subjects
Brief Title: A Drug-Drug Interaction Study in Healthy Volunteers of the Effects of Tucatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONT-380-012
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Drug-drug Interaction
MeSH Terms: interventions — tucatinib; Itraconazole; Rifampin; Gemfibrozil; repaglinide; Tolbutamide; Midazolam; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A (Experimental): Tucatinib plus Itraconazole
  Interventions: Drug: tucatinib; Drug: itraconazole
- Part B (Experimental): Tucatinib plus Rifampin
  Interventions: Drug: tucatinib; Drug: rifampin
- Part C (Experimental): Tucatinib plus Gemfibrozil
  Interventions: Drug: tucatinib; Drug: gemfibrozil
- Part D (Experimental): Tucatinib plus Repaglinide plus Tolbutamide plus Midazolam
  Interventions: Drug: tucatinib; Drug: repaglinide; Drug: tolbutamide; Drug: midazolam
- Part E (Experimental): Tucatinib plus Digoxin
  Interventions: Drug: tucatinib; Drug: digoxin

INTERVENTIONS:
Drug: tucatinib — 300mg dose, orally administered
Drug: itraconazole — 200mg dose
  Arms: Part A
Drug: rifampin — 600mg dose
  Arms: Part B
Drug: gemfibrozil — 600mg tablets
  Arms: Part C
Drug: repaglinide — 1mg dose
  Arms: Part D
Drug: tolbutamide — 500mg dose
  Arms: Part D
Drug: midazolam — 2mg dose
  Arms: Part D
Drug: digoxin — 0.5 mg dose
  Arms: Part E

SUMMARY:
This study is being done to look at how tucatinib could affect the way other drugs work. This study will look at healthy volunteers and how tucatinib affects their liver enzymes. Liver enzymes can change how drugs work in the body. There are 5 parts to this study. Parts A and C are looking at how the body breaks down tucatinib when there are lower levels of certain liver enzymes. Part B is looking at how the body breaks down tucatinib when there are high levels of certain liver and stomach enzymes. Parts D and E are looking at how tucatinib could change the levels of some liver and stomach enzymes in the body. This will help us know more about how tucatinib should be given to patients.

DETAILED DESCRIPTION:
This is a fixed-sequence, drug-drug interaction study of tucatinib conducted in 5 parts in healthy subjects. Part A will evaluate the effect of the strong CYP3A4 inhibitor itraconazole on the pharmacokinetics (PK) of tucatinib. Part B will evaluate the effect of rifampin, a strong inducer of CYP3A4 and CYP2C8, on the PK of tucatinib. Part C will evaluate the effect of the strong CYP2C8 inhibitor gemfibrozil on the PK of tucatinib. Part D will evaluate the effects of tucatinib on the PK of substrate probes of the metabolizing enzymes CYP2C8 (repaglinide), CYP2C9 (tolbutamide), and CYP3A4 (midazolam). Part E will evaluate the effect of tucatinib on the PK of a substrate probe of the transporter P-gp (digoxin). Parts A, B, C, D, and E of the study are independent of one another and do not need to be conducted in a particular order.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 32 kg/m^2
* In good health, determined be no clinically significant findings from medical history, physical examination, and screening evaluations
* Female subjects must be of nonchildbearing potential
* Male subjects must agree to use contraception or must be surgically sterile for at least 90 days prior to enrollment
* Able to understand and sign informed consent form

Exclusion Criteria:

* Any condition affecting drug absorption (including stomach or intestinal surgery)
* Significant history of metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder
* History of hypersensitivity, intolerance, or allergy to any drug compounds, food, or other substance (unless approved by Investigator)
* Participation in a clinical study involving an investigational drug within the past 30 days
* Use or intend to any prescription medications within 28 days prior to check in
* Use of tobacco- or nicotine-containing products within 28 days prior to check in
* History of hyperbilirubinemia
* History of alcoholism or drug abuse within 2 years
* History of regular alcohol consumption exceeding 7 drinks/week for female subjects or 14 drinks/week for male subjects
* Positive hepatitis panel and/or positive human immunodeficiency virus (HIV) test

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time 0 to infinity | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
AUC from time 0 to the time of the last quantifiable concentration | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
Percentage extrapolation in AUC | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
Maximum observed concentration | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
Time of maximum observed concentration | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
Apparent terminal elimination half-life | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide and its M4 metabolite (Part D), tolbutamide and its 4-hydroxytolbutamide metabolite (Part D), midazolam and its 1-hydroxymidazolam metabolite (Part D), and digoxin (Part E)
Apparent total clearance | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide (Part D), tolbutamide (Part D), midazolam (Part D), and digoxin (Part E).
Apparent volume of distribution | Up to 22 days
  PK parameters for tucatinib (Parts A, B, and C); repaglinide (Part D), tolbutamide (Part D), midazolam (Part D), and digoxin (Part E).
Metabolite-to-parent ratio based on AUC | Up to 22 days
  PK parameters for M4 metabolite, 4-hydroxytolbutamide metabolite, and 1-hydroxymidazolam metabolite (Part D only)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 58 days
  Parts A, B, C, D, and E (all)
Incidence of laboratory abnormalities | Up to 58 days
  Parts A, B, C, D, and E (all)
12-lead electrocardiogram (ECG) assessment | Up to 58 days
  PR, RR, QRS, and QT interval. Parts A, B, C, D, and E (all)
Vital signs measurements | Up to 58 days
  Oral temperature. Parts A, B, C, D, and E (all)
Vital signs measurements | Up to 58 days
  Respiratory rate. Parts A, B, C, D, and E (all)
Vital signs measurements | Up to 58 days
  Blood pressure (systolic and diastolic). Parts A, B, C, D, and E (all)
Vital signs measurements | Up to 58 days
  Heart rate. Parts A, B, C, D, and E (all)
Physical examinations | Up to 58 days
  Incidence of AEs resulting from clinically significant findings in examination of general appearance, skin, thorax/lungs, cardiovascular system, and abdomen. Parts A, B, C, D, and E (all)
AUC within a dosing interval | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
AUC from time 0 to infinity | Up to 8 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
AUC from time 0 to the time of the last quantifiable concentration | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Percentage extrapolation in AUC | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Maximum observed concentration | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Time of maximum observed concentration | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Apparent terminal elimination half-life | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Apparent total clearance | Up to 8 days
  PK parameter of tucatinib; Parts D and E only
Apparent total clearance at steady state | Up to 15 days
  PK parameter of tucatinib; Parts D and E only
Apparent volume of distribution | Up to 8 days
  PK parameter of tucatinib; Parts D and E only
Apparent volume of distribution at steady state | Up to 15 days
  PK parameter of tucatinib; Parts D and E only
Accumulation ratio | Up to 15 days
  PK parameters of tucatinib and ONT-993; Parts D and E only
Metabolite-to-parent ratio based on AUC | Up to 15 days
  PK parameter of ONT-993; Parts D and E only

CONTACTS AND LOCATIONS:
Overall Officials: Alex Vo, PhD, Study Director — Seagen Inc.
Locations (2):
- United States (2):
  - Covance Clinical Research Unit, Daytona Beach, Florida
  - Covance Clinical Research Unit, Dallas, Texas

REFERENCES:
- [Derived] Zhang D, Taylor A, Zhao JJ, Endres CJ, Topletz-Erickson A. Population Pharmacokinetic Analysis of Tucatinib in Healthy Participants and Patients with Breast Cancer or Colorectal Cancer. Clin Pharmacokinet. 2024 Oct;63(10):1477-1487. doi: 10.1007/s40262-024-01412-0. Epub 2024 Oct 5. PMID 39368039
- [Derived] Topletz-Erickson A, Lee A, Rustia EL, Sun H, Mayor JG, Abdulrasool LI, Walker L, Endres CJ. Evaluation of Safety and Clinically Relevant Drug-Drug Interactions with Tucatinib in Healthy Volunteers. Clin Pharmacokinet. 2022 Oct;61(10):1417-1426. doi: 10.1007/s40262-022-01144-z. Epub 2022 Aug 6. PMID 35931943